CLINICAL TRIAL: NCT06055153
Title: DV Combined With PD-1 and Platinum-based First-line Treatment in Patients With Locally Advanced or Metastatic HER2 IHC2+/3+ Esophageal Squamous Cell Carcinoma
Brief Title: DV Combined With PD-1 and Platinum-based First-line Treatment in Patients With HER2 IHC2+/3+ ESCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2023-167
Record Dates: First submitted 2023-08-30; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Squamous Carcinoma; HER-2 Protein Overexpression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48+PD-1+platinum-based (Experimental): Dose 1: RC48 2.5mg/kg intravenous infusion, d1 once every 3 weeks;
  Camrelizumab dose: 200mg, intravenous infusion 30-60min, d1 once every 3 weeks;
  Platinum (cisplatin or nedaplatin) : Cisplatin 75mg/m2, added into 500ml 0.9% sodium chloride injection for infusion, hydration and alkalization of -1d, d1, d2, once every 3 weeks; Nedaplatin 75mg/m2 was added to 500ml 0.9% sodium chloride injection, once every 3 weeks.
  Dose 2: rc48 2.0mg/kg, d1, once every 3 weeks; Camrelizumab 200mg, d1 once every 3 weeks; Platinum: Cisplatin 75mg/m2(or nedaplatin 75mg/m2), d1, once every 3 weeks
  Interventions: Drug: RC48+PD-1+platinum-based

INTERVENTIONS:
Drug: RC48+PD-1+platinum-based — Phase I: Three subjects with HER2 overexpression (IHC 2+/3+) were initially enrolled. If dose-limiting toxicity (DLT) was observed in two of the three subjects, the study was continued from dose 1 to dose 2. If ≤1 DLT is observed in 3 subjects, continue to enroll 3 patients, and if ≤2 DLT is observed in 6 subjects, proceed to the second phase. If > 2 cases of DLT are observed in 6 subjects, adjust to dose 2 for phase 2.
  Dose 1: RC48 2.5mg/kg, d1, once every 3 weeks; Camrelizumab 200mg, d1 once every 3 weeks; Platinum: Cisplatin 75mg/m2(or nedaplatin 75mg/m2), d1, once every 3 weeks
  Dose 2: RC48 2.0mg/kg, d1, once every 3 weeks; Camrelizumab 200mg, d1 once every 3 weeks; Platinum: Cisplatin 75mg/m2(or nedaplatin 75mg/m2), d1, once every 3 weeks
  The second stage: sample size expansion stage. RP2D obtained at stage 1 continues to be enrolled in up to 20 patients until disease progression or intolerable toxicity occurs.
  Other Names: Disitamab Vedotin+PD-1+platinum-based

SUMMARY:
This is a single-arm, exploratory clinical study.

DETAILED DESCRIPTION:
This is a single-arm, exploratory clinical study. Aim to explore the safety and efficacy of Vedicetuzumab combined with an immune checkpoint inhibitor (carrellizumab) and platinum-based first-line treatment for locally advanced/metastatic HER2 overexpression (IHC 2+/3+) esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male or female;
2. Patients with locally advanced unresectable, recurrent, or metastatic esophageal cancer were confirmed by imaging examination, and esophageal squamous cell carcinoma was confirmed by histopathology.
3. For those who have received radical therapy and (new) adjuvant therapy, the time of first recurrence or disease progression is greater than 6 months after the end of the last treatment;
4. The HER2 immunohistochemical test was 2+ or 3+;
5. According to the solid tumor Efficacy Evaluation Criteria (RECIST), there should be at least one target lesion that has not received local treatment such as radiotherapy (target lesion located in the previous radiotherapy area can also be selected as a target lesion if it is confirmed to have progressed and meets the RECIST criteria);
6. ECOG score: 0~1;
7. Expected survival≥12 weeks;
8. The function of vital organs met the following requirements (no blood components and cell growth factors were used in the first 2 weeks of enrollment):

   Absolute neutrophil count ≥1.5×109/L Platelet ≥100 × 109/L Hemoglobin ≥90g/L Serum albumin ≥28g/L Bilirubin≤ 1.5 × ULN In the absence of liver metastasis, ALT and AST≤2.5 × ULN; in the presence of liver metastasis, ALT and AST≤5 × ULN Creatinine clearance ≥50ml/min(Cockcroft-Gault); Left ventricular ejection fraction (LVEF) was ≥50% by echocardiography;
9. Fertile female subjects should undergo a urine or serum pregnancy test that proves negative within 72 hours prior to receiving the initial study drug administration and be willing to use an effective method of contraception during the trial period until 3 months after the last dose. For male subjects whose partner is a woman of childbearing age, effective contraception should be used during the trial and within 3 months after the last dose;
10. The subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Other malignancies have been diagnosed within 3 years prior to the first dose, except for effectively treated basal cell carcinoma of the skin, clinical cell carcinoma of the skin, and/or effectively resected cervical and/or breast cancer in situ;
2. There is central nervous system metastasis treatment within one month after stabilization;
3. Have any active autoimmune disease or a history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after normal hormone replacement therapy); Patients with vitiligo or who had complete remission of asthma in childhood and did not require any intervention as adults could be included, but patients with asthma requiring medical intervention with bronchodilators could not be included;
4. suffering from uncontrolled cardiac clinical symptoms or diseases, such as NYHA class II or above heart failure; Unstable angina pectoris; Myocardial infarction within 1 year; Patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
5. Active infection or unexplained fever >38.5℃ occurred during screening or before the first administration of the drug (as determined by the investigator, the subject's fever due to the tumor could be enrolled);
6. Known history or evidence of interstitial lung disease or active non-infectious pneumonia;
7. congenital or acquired immune deficiency (such as HIV infection), active hepatitis B (HBV-DNA≥104/L copy number /ml) or hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the lower detection limit of analytical methods);
8. Known allergic reactions, hypersensitivities or contraindications to macromolecular protein preparations, or to platinum or any component used in preparations there of;
9. Subjects requiring systemic therapy with corticosteroids (>10mg/ day efficacy dose of prednisone) or other immunosuppressants within 14 days prior to initial drug use. In the absence of active autoimmune disease, inhaled or topical steroid and adrenocortical hormone replacement at a therapeutic dose of >10mg/ day of prednisone are permitted;
10. Participate in other clinical studies;
11. Have received live vaccine within 4 weeks prior to the first administration of the drug, and are allowed to receive inactivated virus vaccine for seasonal influenza injection, but are not allowed to receive live attenuated influenza vaccine for nasal administration;
12. Pregnant or lactating women;
13. In the investigator's judgment, the subject has other factors that may lead to the forced termination of the study, such as other serious medical conditions (including mental illness) requiring co-treatment, serious abnormalities in laboratory test values, or family or social factors that may affect the subject's safety or the circumstances of the trial data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase II recommended dose (RP2D) | Up to 28 days
  Defined as maximum tolerated dose or maximum administration dose.
Progression-Free Survival (PFS) | Up to 2 years
  The time between the start of treatment and the onset of disease progression or death

SECONDARY OUTCOMES:
objective response rate (ORR) | Up to 2 years
  The percentage of patients whose tumors have shrunk to a certain amount and remain there for a certain amount of time, including complete response (CR) and partial response (PR) cases

IPD SHARING:
Plan to Share IPD: No